CLINICAL TRIAL: NCT05663125
Title: Safety and Efficacy of LITT Combined With Early Use of Temozolomide for Recurrent Glioblastomas
Brief Title: LITT Combined With Early Use of Temozolomide for Recurrent Glioblastomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dabiao Zhou, MD, Clinical Professor, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-232-01
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Recurrent Glioblastoma
Keywords: GBM; Glioblastoma; LITT; Laser Interstitial Thermal Therapy
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LITT with Early Application of Temozolomide (Experimental): Patients will receive the early use of temozolomide sooner after Laser interstitial thermal therapy (LITT).
  Interventions: Procedure: Laser interstitial thermal therapy; Drug: Temozolomide

INTERVENTIONS:
Procedure: Laser interstitial thermal therapy — Ablation of the tumor will be done by MRI-guided laser interstitial thermal therapy with the assistance of neuro-navigation.
  Other Names: LITT
Drug: Temozolomide — Temozolomide will be administered continuously from the 1st to the 21st day after LITT surgery. The oral dose of temozolomide is 75 mg/m2. And then, it will be given at a routine dose from the second month after surgery.
  Other Names: TMZ

SUMMARY:
This study aims to investigate the safety and efficacy of Laser Interstitial Thermal Therapy (LITT) combined with postoperative early use of temozolomide in treating recurrent glioblastomas.

DETAILED DESCRIPTION:
This is an open-label, non-randomized Phase II study, planning to recruit about ten patients.

The primary objective of this study is to investigate the safety of MRI-guided LITT in combination with the early application of temozolomide.

The secondary outcome is to explore the efficacy of MRI-guided LITT combined with the early use of temozolomide in treating recurrent glioblastomas.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging (PET-MRI) indicates tumor progression or recurrence
2. Patient ≥18 years old
3. The tumor was the first-time recurrence
4. The pathology of the tumor is glioblastoma (IDH wild-type, WHO grade 4)
5. MRI indicated a single tumor or multiple tumors with visual enhancement =<3cm
6. Maximum tumor diameter: single tumor =<3cm; Multiple tumors, targeted lesion =<3cm
7. Single tumor or one of the multiple tumor lesions involved deep functional areas such as the insula lobe or thalamus
8. KPS score >=60 within 30 days before treatment
9. No serious liver or kidney dysfunction
10. Patients must be able to understand how to sign the informed consent document

Exclusion Criteria:

1. The tumor crossed the midline or involved bilateral cerebral hemispheres
2. Inability to perform MRI examination or intolerance to MRI contrast agent
3. There is an active infection of the patient
4. The patient had abnormal coagulation function
5. Imaging before treatment indicated signs of cerebral hernia or midline displacement > 1.0cm
6. The patient received radiotherapy, chemotherapy (including immunotherapy), or other therapeutic measures after tumor recurrence
7. Patients who have participated in clinical trials of any other drug or medical device within three months of the screening.
8. KPS score =<50 points

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From Day 1 throughout the study until 3 months
  To complete protocol treatment without undue treatment-related acute toxicity in recurrent glioblastoma patients undergoing LITT followed by early use of temozolomide.

SECONDARY OUTCOMES:
Time to Progression (TTP) | 12 months
  TTP, defined as time from LITT to recorded tumor progression
Overall survival (OS) | 18 months
  OS, defined as time from diagnosis to death

CONTACTS AND LOCATIONS:
Overall Officials: Dabiao Zhou, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No